CLINICAL TRIAL: NCT04754880
Title: The Relationship Between Oxidative Stress Markers and Presence of Chronic Total Occlusion in Coronary Artery Disease
Brief Title: Coronary Chronic Total Occlusion and Oxidative Balance
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ekrem Aksu, Assis. Prof. MD, Kahramanmaras Sutcu Imam University
Other Study IDs: 14.10.2020-2020/19/16
Record Dates: First submitted 2021-01-30; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Progression of Atherosclerotic Plaque; Coronary Artery Disease
Keywords: chronic total occlusion, oxidative balance, stable coronary artery disease, vitamin A, vitamin C, vitamin C/vitamin A ratio.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-CTO: This group was defined as no chronic obstruction, except for non-critical stenosis, who underwent coronary angiography with the diagnosis of stable angina pectoris.
  Interventions: Diagnostic Test: Comparison of oxidative and antioxidative markers between groups
- CTO: This group was defined as the presence of complete occlusion in one artery and no critical lesions (> 50%) in the other arteries undergoing coronary angiography with the diagnosis of stable angina pectoris.
  Interventions: Diagnostic Test: Comparison of oxidative and antioxidative markers between groups

INTERVENTIONS:
Diagnostic Test: Comparison of oxidative and antioxidative markers between groups — Oxidant and anti-oxidant markers

SUMMARY:
The presence of chronic blockage of coronary arteries, which we may accept as the terminal point of atherosclerotic coronary artery disease, is closely associated with a poor prognosis. The Discovery of markers that may distinguish patients with a high risk of chronic total occlusion development among patients monitored with the diagnosis of stable coronary artery disease may be important for being able to reduce the increased mortality and morbidity rates.

Oxidative stress status may be one of the markers that play a role in and/or show the development of chronic total occlusion. It was reported that it has a role in the progression, erosion, and instability of atherosclerotic plaques in coronary arteries. To the best of our knowledge, the relationship between chronic total occlusion development and oxidative stress status in stable coronary artery disease has not been studied.

This study investigated the relationships in the oxidative stress status evaluated over TAS, TOS, OSI, Thiol/Disulfide Homeostasis, and antioxidative vitamin levels and possible differences in patients with noncritical coronary artery disease and those with chronic total occlusion.

DETAILED DESCRIPTION:
Chronic total occlusion (CTO) is defined as the complete blockage of the coronary artery characterized by a TIMI 0 flow present for at least 3 months. The presence of chronic blockage of coronary arteries, which we may accept as the terminal point of atherosclerotic coronary artery disease, is closely associated with a poor prognosis. In coronary angiography tests conducted due to stable angina pectoris, it was observed that the incidence of chronic total occlusion varied in the range of 15-30%. Moreover, its actual incidence in society is unknown as it is generally asymptomatic. The Discovery of markers that may distinguish patients with a high risk of chronic total occlusion development among patients monitored with the diagnosis of stable coronary artery disease may be important for being able to reduce the increased mortality and morbidity rates.

Oxidative stress status may be one of the markers that play a role in and/or show the development of chronic total occlusion. Reactive oxygen species which show an increase in the case of oxidative stress emerging by increased production of oxidants on the cellular level or a reduced antioxidant system result in disorders on the tissue and organ levels as a result of the damages they induce on DNA, protein, and lipid structures. It was reported that it has a role in the progression, erosion, and instability of atherosclerotic plaques in coronary arteries. Furthermore, the relationship between oxidative stress and the progression of atherosclerosis in coronary arteries has been usually studied in acute coronary syndrome patients. To the best of our knowledge, the relationship between chronic total occlusion development and oxidative stress status in stable coronary artery disease has not been studied.

This study investigated the relationships in the oxidative stress status evaluated over TAS, TOS, OSI, Thiol/Disulfide Homeostasis, and antioxidative vitamin levels and possible differences in patients with noncritical coronary artery disease and those with chronic total occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Those who underwent coronary angiography with the diagnosis of stable coronary artery disease
* Elder than 18 years
* Patients who were not have the exclusion criterias

Exclusion Criteria:

* Being under the age of 18,
* Unstable angina pectoris,
* Left ventricular systolic dysfunction (Ejection fraction <50),
* Severe anemia
* pregnancy,
* History of congenital heart disease,
* Thyroid disorders,
* Sepsis,
* Malignancy,
* Chronic hematological disease,
* Malnutrition,
* Collagen tissue disease,
* Obesity (The Body Mass Index >(BMI 30 kg/m2) ,
* moderate to severe liver failure,
* Renal deficiency (Glomerular filtration rate <60 ml/min/1.73m2),
* Severe heart valve disease,
* Slectrolyte disorders,
* Receiving multivitamin and antioxidant supplementation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study consecutively included 29 patients who received coronary angiography with the diagnosis of stable angina pectoris and had a presence of total occlusion in one artery and no critical lesion (>50%) in other arteries in the patient group.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between oxidative balance and chronic total occlusion in stable coronary artery disease | 24 months
  Serum Total thiol (μmol / L), Native thiol (μmol / L), Disulfide (μmol / L), Total oxidant status (TOS) (umol/L), Total antioxidant status (TAS) (mmol/L), Oxidative stress index (TOS/TAS), Vitamin A, ng/ml, Vitamin C (ng/ml), Vitamin C / Vitamin A Ratio will be measured and the correlation of these markers with chronic total occlusion of the coronary artery will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ekrem Aksu, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Lesiak M, Cugowska M, Araszkiewicz A, Grygier M, Pyda M, Skorupski W, Mitkowski P, Lanocha M, Grajek S. Impact of the presence of chronically occluded coronary artery on long-term prognosis of patients with acute ST-segment elevation myocardial infarction. Cardiol J. 2017;24(2):117-124. doi: 10.5603/CJ.a2016.0112. Epub 2016 Dec 2. PMID 27910082
- [Background] Kahn JK. Angiographic suitability for catheter revascularization of total coronary occlusions in patients from a community hospital setting. Am Heart J. 1993 Sep;126(3 Pt 1):561-4. doi: 10.1016/0002-8703(93)90404-w. PMID 8362709
- [Background] Gulcin I. Antioxidants and antioxidant methods: an updated overview. Arch Toxicol. 2020 Mar;94(3):651-715. doi: 10.1007/s00204-020-02689-3. Epub 2020 Mar 16. PMID 32180036
- [Background] Increased thiol/disulphide ratio in patients with ST elevation-acute coronary syndromes. Cukurova Medical Journal 2019;44(1):20-25.
- [Background] Borekci A, Gur M, Turkoglu C, Selek S, Baykan AO, Seker T, Harbalioglu H, Ozaltun B, Makca I, Aksoy N, Gozukara Y, Cayli M. Oxidative Stress and Spontaneous Reperfusion of Infarct-Related Artery in Patients With ST-Segment Elevation Myocardial Infarction. Clin Appl Thromb Hemost. 2016 Mar;22(2):171-7. doi: 10.1177/1076029614546329. Epub 2014 Aug 12. PMID 25115763
- [Background] Gensini GG. A more meaningful scoring system for determining the severity of coronary heart disease. Am J Cardiol. 1983 Feb;51(3):606. doi: 10.1016/s0002-9149(83)80105-2. No abstract available. PMID 6823874